CLINICAL TRIAL: NCT00639496
Title: Idiopathic Pulmonary Fibrosis International Group Exploring NAC I Annual Study of the Effects of High-dose N-acetylcysteine (NAC) in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study of the Effects of High-dose N-acetylcysteine (NAC) in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: IFIGENIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7112LAMC01
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2008-03

CONDITIONS: Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patients taking NAC 600 mg t.i.d.
  Interventions: Drug: n-acetylcysteine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: n-acetylcysteine — 600 mg x 3, for 12 months
  Other Names: Flumucil
  Arms: 1
Drug: placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether NAC added to prednisone, and azathioprine has a better effect on lung function, radiology and clinical condition than placebo + prednisone in combination with azathioprine after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF according to the International Consensus Statement
* Bronchoalveolar lavage (BAL) showing no features to support an alternative diagnosis.
* Patients in whom it was possible to determine single breath DLco.
* Patients with newly or previously diagnosed IPF, in whom it was clinically justified to use the standardised regimen azathioprine plus prednisone

Exclusion Criteria:

* Known intolerance to N-Acetylcysteine.
* Patients with respiratory infections at study entry should be excluded until the infections have been treated successfully (VC and Dlco comparable with the values before the infection).
* Patients with pre-existing disease that interferes with the evaluation of IPF: extensive old TBC lesions, significant bronchiectasis, moderate or severe COPD.
* Patients with malignancy in the last 5 years. If the patient had a malignancy in the past and is free of malignancy for more than five years, the patient is regarded as healed.
* Patients with heart failure.
* Patients with hepatic function abnormalities contraindicating the use of azathioprine (i.e. clinically significant abnormalities of PTT and/or GGT).
* Patients with a renal clearance < 10ml/min and/or hematuria and/or proteinuria of collagen vascular disease origin. A renal clearance is only performed in the presence of an abnormal serum creatinine and/or serum urea level.
* Patients who are artificially ventilated.
* Prednisone at a dose > 0.5 mg/kg/day (or other glucocorticoids such as triamcinolone, dexamethasone or methylprednisolone at an equivalent dose) or azathioprine at a dose > 2 mg/kg/day during the last month prior to inclusion.
* Use of other immunosuppressives (such as cyclophosphamide and colchicine) is not allowed in the last month and for the duration of the trial.
* Any form of anticancer therapy or methotrexate are not allowed when used for more than 1 week in the past and for the duration of the trial.
* Amiodarone or nitrofurantoin are not allowed in the last 5 years, when used for more than 1 week in the past and for the duration of the trial.
* Allopurinol, oxypurinol, thiopurinol, anti-oxidants (e.g. vitamin E) or glutathione supplements are not allowed in the last month and during the trial.
* The use of interferon or other antifibrotics (e.g. pirfenidone) is not allowed in the past and during the study.
* The use of NAC therapy at a dosage of more than 600 mg/day is not allowed in the last 3 years for a total period of more than 3 months.
* Patients suffering or having suffered from documented active ulcer within the last 3 years.
* Patients in whom the standardised treatment regimen is contraindicated or not justified.
* Pregnancy.
* Known or suspected drug or alcohol abuse.
* Patients on other investigational compounds or participating in clinical trials on investigational compounds within the last 3 months.
* Patients expected to be non-compliant in taking the medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2000-03; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Vital capacity (VC) and diffusion capacity for CO (DLCO) | at 6 and 12 months

SECONDARY OUTCOMES:
clinical, radiologic and physiologic (CRP)-score | at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Demedts, MD, Study Chair — U.Z.-Gasthuisberg, Leuven, Belgium
Locations (7):
- U.Z. Ghent, Ghent, Belgium
- Hôpital A. Calmette, Lille, France
- Klinikum Grosshadern, Munich, Germany
- U.O. di Pneumologia-Ospedale, Arezzo, Italy
- Stichting St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Hospital Universitario Virgen del Rocío, Seville, Spain
- The University of Edinburgh-Medical School, Edinburgh, United Kingdom

REFERENCES:
- [Result] Demedts M, Behr J, Buhl R, Costabel U, Dekhuijzen R, Jansen HM, MacNee W, Thomeer M, Wallaert B, Laurent F, Nicholson AG, Verbeken EK, Verschakelen J, Flower CD, Capron F, Petruzzelli S, De Vuyst P, van den Bosch JM, Rodriguez-Becerra E, Corvasce G, Lankhorst I, Sardina M, Montanari M; IFIGENIA Study Group. High-dose acetylcysteine in idiopathic pulmonary fibrosis. N Engl J Med. 2005 Nov 24;353(21):2229-42. doi: 10.1056/NEJMoa042976. PMID 16306520
- [Derived] Behr J, Demedts M, Buhl R, Costabel U, Dekhuijzen RP, Jansen HM, MacNee W, Thomeer M, Wallaert B, Laurent F, Nicholson AG, Verbeken EK, Verschakelen J, Flower CD, Petruzzelli S, De Vuyst P, van den Bosch JM, Rodriguez-Becerra E, Lankhorst I, Sardina M, Boissard G; IFIGENIA study group. Lung function in idiopathic pulmonary fibrosis--extended analyses of the IFIGENIA trial. Respir Res. 2009 Oct 27;10(1):101. doi: 10.1186/1465-9921-10-101. PMID 19860915